CLINICAL TRIAL: NCT01181323
Title: A Randomized, Double-Blind Trial, Comparing the Safety in Mothers and Their Infants and Immunogenicity in Mothers of Live Attenuated Influenza Vaccine (LAIV) to Inactivated Trivalent Influenza Vaccine (TIV) When Administered to Breast Feeding Women
Brief Title: Post-Partum Immunization With Live Attenuated Influenza Vaccine (LAIV) or Trivalent Influenza Vaccine (TIV) in Post-Partum Breast Feeding Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0007; HHSN272200800006C
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2013-04

CONDITIONS: Influenza
Keywords: influenza, vaccine, breastfeeding, post-partum women, infant, LAIV, TIV, parent protocol
MeSH Terms: conditions — Influenza, Human; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Group 1: LAIV (Experimental): 0.2 ml of Live attenuated influenza vaccine (LAIV), Flumist® given intranasally (IN) and 0.5 ml of placebo given intramuscularly (IM) injection administered to 120 maternal subjects.
  Interventions: Biological: Cold-adapted live attenuated influenza virus vaccine, trivalent; Other: Placebo
- Group 2: TIV (Experimental): 0.5 ml of Inactivated Trivalent Influenza Vaccine (TIV), Fluzone® given intramuscularly (IM) and 0.2 ml of placebo given intranasally (IN) administered to 120 maternal subjects.
  Interventions: Other: Placebo; Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Other: Placebo — 0.2 ml of Intranasal placebo study product (using sucrose phosphate placebo filled sprayers), will be administered to maternal subjects.
  Arms: Group 2: TIV
Biological: Cold-adapted live attenuated influenza virus vaccine, trivalent — Licensed product formulated for the 2011-2012 or 2012-2013 influenza season. Standard dose LAIV (Flumist®) 0.1 ml administered to maternal subjects intranasally in each nostril for a total of 0.2 mL.
  Arms: Group 1: LAIV
Other: Placebo — 0.5 ml of Sterile saline (0.9 percent Sodium Chloride for injection), administered IM to maternal subjects.
  Arms: Group 1: LAIV
Biological: Trivalent inactivated influenza vaccine — Preservative free, licensed product formulated for the 2011-2012 or 2012-2013 influenza season. Standard dose of TIV (Fluzone®) 0.5 ml administered to maternal subjects, IM in the deltoid.
  Arms: Group 2: TIV

SUMMARY:
The purpose of this research study is to learn more about the safety of 2 licensed flu vaccines, nasal spray and flu vaccine shot, in mothers and their infants, when given to women who are breastfeeding and to compare the immune response (body's defense against foreign substances) of breastfeeding mothers, who receive intranasal flu vaccine, with breastfeeding mothers receiving the flu vaccine shot. Healthy women (240 volunteers, 28-120 days post delivery) who plan to breastfeed through 28 days post vaccination and who have not received influenza vaccine for the influenza season for which they are being enrolled, will be assigned by chance to 1 of the 2 vaccines in the following manner: flu vaccine nasal spray and a placebo (inactive substance) shot or a flu vaccine shot and a placebo nasal spray. Study procedures include: nasal swabs, blood samples, and completion of memory aids. Participants will be involved in this United States based study for about 6 months.

DETAILED DESCRIPTION:
Due to limited data available on the safety and immune response to live attenuated influenza vaccine (LAIV) in breast-feeding women and the lack of information on the induction of immunoglobulin (Ig) A and IgG against influenza virus in breast milk, this study compares the safety in mothers and their infants and immunogenicity in mothers of standard dose inactivated trivalent influenza vaccine (TIV) and LAIV when administered between 28-120 days of delivery in breastfeeding women. This is a multi-site, randomized, double-blinded trial in 240 post-partum breastfeeding women, 18-49 years of age and their infants. Once enrolled, a blood sample and a breast milk sample will be collected. Nasal swabs will be obtained and targeted physical examinations (TPE) will be conducted from mother and infant, if indicated. Each subject will receive either a single intramuscular (IM) 0.5 milliliter (mL) dose of TIV and 0.2 mL of placebo administered intranasally, or 0.2 mL intranasal dose of LAIV and 0.5 mL of placebo administered IM. All subjects will maintain a memory aid recording oral temperature, and systemic and local adverse events (AEs) for 8 days after study products have been administered. Approximately day 2 and 8 all subjects will return to the clinic for collection of breast milk samples and nasal swabs (mother and infant) and the memory aid will be reviewed. Approximately Day 28 after vaccination, all subjects will return to the clinic for breast milk and a blood sampling. During the time between vaccination and the day 28 visit, if mother or infant has an influenza-like illness (ILI), a clinic visit may be required within 72 hours of illness onset. The clinic visit will be required for any illness that meets the Centers for Disease Control and Prevention's definition of an ILI for the mother. Investigator discretion will discern if an illness in the infant requires an ILI visit. Any respiratory or gastrointestinal (GI) serious adverse event (SAE) in the infant will also require a clinic visit. If the mother has an ILI, nasal swabs will be collected on her, and samples from the infant (if possible). If the infant has an ILI, nasal swabs will be collected on both the mother and infant. At approximately Day 42 after vaccination, all subjects will have a phone call for assessment of any medically attended GI or respiratory illness in the infant from Day 29-42. Approximately 6 months after vaccination all subjects will have a phone call for assessment of any SAEs in the subject or the infant since Day 42. SAE data and new onset chronic medical conditions in the mother will be collected from Day 0-180. At all study visits, subjects will be asked about acute, temporary breast diseases (mastitis, abscesses) and any changes in breastfeeding, i.e., interruption and if so, how long (in weeks). Subjects will report information on current breast milk consumption by infant. Unsolicited non-serious AE data will be captured Day 0-28. Respiratory and GI AEs will be captured for the infant from Day 28-42. SAE data will be captured from Day 0-180 for both mother and infant. Blood samples will be tested for hemagglutination inhibition (HAI), IgG, and IgA as measured by enzyme linked-immunosorbent assay (ELISA). Breast milk samples will be assayed for IgA and IgG antibodies by ELISA. Breast milk and nasal swabs will also be tested for LAIV. Parent protocol to sub-study 11-0048.

ELIGIBILITY:
Inclusion Criteria:

Maternal Subject

* Women age 18-49 years of age (inclusive) within 28-120 days of delivery.
* Is in good health, as determined by vital signs (heart rate </=100 beats per minute (bpm); blood pressure: systolic <150 mm Hg; diastolic <90 mm Hg; oral temperature <100.0 degrees Fahrenheit), medical history and a targeted physical examination if indicated based on medical history.
* Willing and capable of providing written informed consent for herself and infant.
* Available for entire study duration, clinic visits and phone calls.
* Planning on breast feeding from time of vaccination through 28 days post-vaccination. Breast milk must be at least one half of the source of the infant's feeding.
* Willing to practice adequate contraception for at least 28 days after receipt of study vaccine if not surgically sterile via post-partum tubal ligation, bilateral oophorectomy or hysterectomy. Adequate contraception may include, but is not limited to, abstinence, monogamous relationship with a vasectomized partner, barrier methods such as condoms or diaphragms with spermicides, or licensed hormonal methods that are compatible with breastfeeding an infant.
* May be reached by any IRB-approved form of communication during study period. May include telephone, email, web based, social media, and/or text messaging, based on specific local IRB recommendations.
* Agree to sign a medical release for herself and her infant (if needed) so that study personnel may obtain medical information about her or her infant's health.

Infant The infant(s) should be in good health as assessed by medical history, interview, rectal temperature and a targeted physical examination based on medical history.

* Infant born greater than or equal to 36 weeks gestation.
* Successful receipt of breast milk for at least two days prior to enrollment. Breast milk must be at least one half of the source of feeding, i.e., some supplementation is acceptable.

Exclusion Criteria:

Maternal Subject

* History of receipt of licensed influenza vaccine for the current influenza season. (If enrolled in 2011-2012 season [October 2011 - February 2012], subject must not have received 2011-2012 influenza vaccine. If enrolled in the 2012-2013 season [July 2012 or later], subject must not have received 2012-2013 influenza vaccine).
* History of previous participation in this study.
* Known allergy to eggs, egg proteins or other components in the vaccines (i.e. formaldehyde, polyethylene glycol, p-isooctylphenyl ether, sucrose, gelatin, polysorbate 80, gentamicin, arginine, sodium phosphate, sodium chloride, octylphenol ethoxylate, EDTA).
* If enrolled in the 2011-2012 season, known or suspected latex allergy. For the 2012-2013 season, known or suspected latex allergy is not a reason for exclusion.
* History of severe reactions following immunization with contemporary influenza virus vaccines.
* Received any other licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to vaccination in this study, or expects to receive a licensed vaccine during the 28 days after vaccination in this study.
* Received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 28 days prior to vaccination in this study, or expects to receive an experimental/investigational agent within the study time period (180 days after vaccination in this study).
* Received antiviral agent against influenza A and/or B within 48 hours prior to vaccination in this study. Antiviral agents should not be administered until 2 weeks after vaccination in this study unless medically necessary.
* A moderate to severe acute illness and/or an oral temperature >/= 100.0 F, within 72 hr prior to vaccination. (This may result in a temporary delay of vaccination).
* Immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Active neoplastic disease or a history of any hematologic malignancy (cancers of blood or bone marrow) or current bleeding or blood clotting disorder.
* Current diagnosis of asthma.
* History of asthma, wheezing, or bronchospasm in the last 5 years.
* Long term (at least 14 days of prednisone 2 mg/kg or equivalent other glucocorticoid) use of oral or parenteral steroids, high-dose inhaled steroids (>800 microgram/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (topical steroids are allowed).
* Use of intranasal steroids within 14 days prior to vaccination in this study or within 14 days after receipt of study vaccine.
* Use of intranasal products within 6 hours prior to vaccination in this study or expects to use intranasal products within 6 hours post study vaccination.
* History of receiving immunoglobulin or other blood product (with exception of RhoGAM) within the 3 months prior to vaccination in this study.
* Diagnosis of a current and uncontrolled major psychiatric disorder.
* Has been hospitalized within the past 10 years for psychiatric illness, suicide attempt, or confinement for danger to self or others.
* The subject is receiving listed psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* The subject is receiving medications contraindicated with breast feeding.
* Known active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
* An active neurological (such as, but not limited to seizure disorder), auto-immune or vascular disease.
* Active breast infection or breast abscess. (Study vaccination will be delayed until this breast infection or breast abscess has been treated and is resolved.)
* History of frequent epistaxis (nose bleeds).
* History of alcohol or drug abuse in the 1 year prior to enrollment.
* History of Guillain-Barré syndrome.
* Any known immunocompromised family member/household contact (such as active cancer, lupus, inflammatory bowel disease, HIV infection, or receipt of an organ or bone marrow transplant).
* Has an acute or chronic medical condition that, in the opinion of the investigator would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver, lung or heart disease, chronic anemia, metabolic disorders such as diabetes (resolved gestational diabetes is acceptable), significant renal disease, transplant recipients).
* Pregnant or planning to become pregnant during the 28 days after receipt of study vaccine.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Infant

* Major congenital malformations.
* Syndromes that affect breastfeeding.
* Progressive neurological disease or a history of any seizure.
* Chronic lung disease or oxygen requirement for heart disease.
* History of bronchopulmonary dysplasia, wheezing, reactive airway disease, hospitalization for respiratory illness, or use of bronchodilators.
* Any receipt of glucocorticoids.
* Immunodeficiency disease or use of immunosuppressive therapy including perinatal exposure to or infection with HIV, or known infection with hepatitis B or hepatitis C.
* Received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 28 days prior to this study, or expects to receive an experimental/investigational agent within the study time period (180 days after mother's vaccination in this study).
* A moderate to severe acute illness and/or a rectal temperature greater than or equal to 100.0 F (37.8 C), within 72 hours prior to mother's vaccination (This may result in a temporary delay of vaccination in mother).
* Received any licensed vaccines within 7 days prior to mother's vaccination in this study, or expects to receive a licensed vaccine during the 10 days after mother's vaccination in this study (This may result in a temporary delay of vaccination in mother).
* History of documented laboratory-confirmed influenza infection.
* Receipt of blood or blood products.
* Have a condition that may place the infant at an unacceptable risk of injury or would make it difficult for the infant to meet the requirements of the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Washington Hospital Center - Obstetrics and Gynecology, Washington D.C., District of Columbia
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Translational Medicine Institute - Clinical Vaccine Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Group Health Research Institute - Seattle, Seattle, Washington

REFERENCES:
- [Derived] Brady RC, Jackson LA, Frey SE, Shane AL, Walter EB, Swamy GK, Schlaudecker EP, Szefer E, Wolff M, McNeal MM, Bernstein DI, Steinhoff MC. Randomized trial comparing the safety and antibody responses to live attenuated versus inactivated influenza vaccine when administered to breastfeeding women. Vaccine. 2018 Jul 25;36(31):4663-4671. doi: 10.1016/j.vaccine.2018.06.036. Epub 2018 Jun 28. PMID 29961606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy post-partum women recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 6Sep2011 and 31Oct2012
Pre-assignment Details: Maternal participants and their infants were enrolled separately in the study for the purposes of data collection, analysis and reporting. For baseline measures, adverse events, and outcome measures as appropriate, the infants are defined as their own arms of the study based on the study product the mother received.
Groups:
- Maternal LAIV: Healthy women who planned to breast feed through 28 days post vaccination received 0.2 mL of licensed live attenuated influenza vaccine (LAIV), Flumist®, intranasally, and 0.5 ml of sterile saline placebo by intramuscular injection
- Maternal TIV: Healthy women who planned to breast feed for 28 days post vaccination received 0.5 mL licensed seasonal trivalent influenza vaccine (TIV) by intramuscular injection, Fluzone®, by intramuscular injection, and 0.2 mL sucrose phosphate placebo intranasally.
- Infant LAIV: Infants of women enrolled to receive LAIV were enrolled separately in the protocol to be followed for safety outcomes.
- Infant TIV: Infants of women enrolled to receive TIV were enrolled separately in the protocol to be followed for safety outcomes.
Period: Overall Study
Arm/Group | Maternal LAIV | Maternal TIV | Infant LAIV | Infant TIV
Started | 124 | 124 | 124 | 125
Completed | 123 | 121 | 123 | 122
Not Completed | 1 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled subjects are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal LAIV | Maternal TIV | Infant LAIV | Infant TIV | Total
Number analyzed (Participants) | 124 | 124 | 124 | 125 | 497
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 124 | 125 | 249
  Between 18 and 65 years | 124 | 124 | 0 | 0 | 248
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 124 | 61 | 62 | 371
  Male | 0 | 0 | 63 | 63 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 2 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 1 | 3
  Black or African American | 13 | 11 | 10 | 11 | 45
  White | 98 | 98 | 95 | 93 | 384
  More than one race | 6 | 9 | 17 | 17 | 49
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 10 | 6 | 23
  Not Hispanic or Latino | 118 | 123 | 114 | 119 | 474
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 124 | 124 | 124 | 125 | 497

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation thereof; was a congenital anomaly/birth defect; or may have jeopardized the participant, or required intervention to prevent one of the outcomes, regardless of relationship to study product or study participation.
Time Frame: Day 0 to Day 180 post vaccination
Population: All enrolled participants are included in the analysis population for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV | Maternal TIV | Infant LAIV | Infant TIV
Number analyzed (Participants) | 124 | 124 | 124 | 125
participants | 1 | 0 | 2 | 1

2. Primary Outcome: Number of Participants Reporting New Onset Chronic Medical Conditions
Description: New onset chronic medical condition was defined as any new ICD-10 diagnosis for a participant that was expected to continue for at least 6 months and require continued health care intervention. ICD-10 = International Statistical Classification of Diseases and Related Health Problems, 10th revision. Maternal participants were asked at each visit through 180 days after enrollment if they or their infants had any new diagnosis.
Time Frame: Day 0 to Day 180 post vaccination
Population: All enrolled participants are included in the analysis population for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV | Maternal TIV | Infant LAIV | Infant TIV
Number analyzed (Participants) | 124 | 124 | 124 | 125
participants | 1 | 1 | 3 | 4

3. Primary Outcome: Number of Infant Participants Reporting Solicited Systemic Adverse Events Within 11 Days of Maternal Vaccination
Description: Maternal participants maintained a memory aid to record daily the occurrence in their infants of systemic adverse events of fever (defined as rectal temperature 37.8 degrees Celsius or greater), drowsiness, irritability/fussiness, loss of appetite, nasal congestion, difficulty breathing, runny nose, and cough for 11 days (Day 0-10) after maternal vaccination based on protocol-defined grading (none, mild, moderate or severe) for each symptom. Rectal temperature was measured once daily. Participants are counted if they were reported as experiencing the symptom at any severity on any of the 11 days.
Time Frame: Day 0 to Day 10 post vaccination
Measure: Number; unit: participants
Arm/Group | Infant LAIV | Infant TIV
Number analyzed (Participants) | 124 | 125
participants
  Fever | 28 | 23
  Drowsiness | 42 | 33
  Irritability/fussiness | 74 | 56
  Loss of appetite | 20 | 14
  Nasal congestion | 54 | 54
  Difficulty breathing | 12 | 7
  Runny nose | 18 | 30
  Cough | 15 | 18

4. Primary Outcome: Number of Participating Reporting Non-serious Unsolicited Adverse Events Related to Vaccination Within 28 Days of Maternal Vaccination
Description: Adverse events (AE) for this protocol used the International Conference on Harmonization (ICH) guideline E6 definition of AE, any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product regardless of its causal relationship to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product. Related was defined as a reasonable possibility that the study product caused the AE. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event. Non-serious AEs were those that did not meet the definition of serious (see Outcome Measure 1). Maternal participants were queried at each visit through 28 days after vaccination for the occurrence of any AE for her or the infant separately from the pre-defined solicited symptoms.
Time Frame: Day 0 to Day 28 post vaccination
Population: All enrolled participants are included in the analysis population for this outcome measure
Measure: Number; unit: participants
Arm/Group | Maternal LAIV | Maternal TIV | Infant LAIV | Infant TIV
Number analyzed (Participants) | 124 | 124 | 124 | 125
participants | 6 | 3 | 5 | 8

5. Primary Outcome: Breast Milk ELISA IgA and IgG Geometric Mean Titers (GMT) to Each of the Vaccine Influenza Strains
Description: Breast milk was collected at Day 0 prior to vaccination and again at 28 days following vaccination for testing in IgA and IgG ELISA Assays. The ELISA assay was conducted with the antigens in the 2011-2012 seasonal influenza vaccine, A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008, those in the 2012-2013 seasonal influenza vaccine, A/Victoria/361/2011 and B/Wisconsin/1/2010, and the antigen in both seasons's vaccine, A/California/7/2009 (H1N1). The lower limit of detection is 5.82 units/mL for IgA and 2.56 units/mL for IgG. Titers below the limit of detection were reported as one-half the limit of detection.
Time Frame: Day 0 and 28 post vaccination
Population: All enrolled maternal participants are included in this analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: units/mL
Groups:
- Maternal LAIV 2011-2012: Healthy women who planned to breast feed through 28 days post vaccination received 0.2 mL of licensed live attenuated influenza vaccine (LAIV), Flumist®, intranasally in the 2011-2012 season
- Maternal LAIV 2012-2013: Healthy women who planned to breast feed through 28 days post vaccination received 0.2 mL of licensed live attenuated influenza vaccine (LAIV), Flumist®, intranasally in the 2012-2013 season
- Maternal TIV 2011-2012: Healthy women who planned to breast feed for 28 days post vaccination received 0.5 mL licensed seasonal trivalent influenza vaccine (TIV) by intramuscular injection, Fluzone®, by intramuscular injection in the 2011-2012 season
- Maternal TIV 2012-2013: Healthy women who planned to breast feed for 28 days post vaccination received 0.5 mL licensed seasonal trivalent influenza vaccine (TIV) by intramuscular injection, Fluzone®, by intramuscular injection in the 2012-2013 season
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Maternal TIV 2011-2012 | Maternal TIV 2012-2013
Number analyzed (Participants) | 76 | 48 | 74 | 50
units/mL
  Day 0 IgA to A/California/7/2009 (H1N1) | 8.8 [6.6 to 11.7] | 8.6 [6.1 to 12.2] | 8.7 [6.3 to 12.0] | 7.5 [5.1 to 11.0]
  Day 28 IgA to A/California/7/2009 (H1N1) | 9.0 [6.6 to 12.4] | 10.5 [7.5 to 14.7] | 23.2 [15.2 to 35.4] | 10.8 [7.4 to 15.8]
  Day 0 IgA to A/Perth/16/2009 (H3N2) | 22.9 [17.1 to 30.6] | 32.8 [24.4 to 44.2] | 20.9 [15.5 to 28.1] | 23.8 [15.7 to 36.0]
  Day 28 IgA to A/Perth/16/2009 (H3N2) | 29.3 [21.3 to 40.2] | 50.8 [37.1 to 69.4] | 44.2 [31.6 to 61.8] | 38.9 [25.0 to 60.4]
  Day 0 IgA to A/Victoria/361/2011 (H3N2) | 22.5 [16.7 to 30.4] | 33.9 [23.6 to 48.7] | 22.7 [16.8 to 30.7] | 24.7 [16.6 to 36.7]
  Day 28 IgA to A/Victoria/361/2011 (H3N2) | 28.5 [20.7 to 39.1] | 51.8 [37.9 to 70.9] | 46.0 [32.7 to 64.5] | 44.2 [28.3 to 69.0]
  Day 0 IgA to B/Brisbane/60/2008 | 17.1 [13.4 to 21.8] | 15.9 [11.1 to 22.7] | 12.9 [9.8 to 16.8] | 15.1 [10.9 to 20.8]
  Day 28 IgA to B/Brisbane/60/2008 | 22.9 [17.2 to 30.3] | 22.0 [15.0 to 32.3] | 23.9 [17.4 to 32.8] | 23.4 [16.5 to 33.4]
  Day 0 IgA to B/Wisconsin/1/2010 | 8.2 [6.4 to 10.6] | 10.0 [7.1 to 14.1] | 8.3 [6.3 to 10.8] | 7.5 [5.6 to 10.1]
  Day 28 IgA to B/Wisconsin/1/2010 | 10.6 [7.9 to 14.1] | 15.3 [9.9 to 23.5] | 10.7 [7.9 to 14.6] | 21.2 [13.6 to 33.1]
  Day 0 IgG to A/California/7/2009 (H1N1) | 1.6 [1.4 to 1.8] | 1.6 [1.3 to 1.9] | 1.7 [1.5 to 2.0] | 1.7 [1.4 to 2.1]
  Day 28 IgG to A/California/7/2009 (H1N1) | 1.6 [1.4 to 1.8] | 1.6 [1.4 to 1.9] | 5.0 [3.7 to 6.7] | 2.9 [2.2 to 3.9]
  Day 0 IgG to A/Perth/16/2009 (H3N2) | 2.4 [2.0 to 2.9] | 2.6 [2.1 to 3.4] | 2.1 [1.7 to 2.5] | 2.7 [2.0 to 3.5]
  Day 28 IgG to A/Perth/16/2009 (H3N2) | 2.3 [1.9 to 2.9] | 2.9 [2.3 to 3.8] | 5.5 [4.3 to 7.2] | 6.7 [5.0 to 8.9]
  Day 0 IgG to A/Victoria/361/2011 (H3N2) | 2.6 [2.1 to 3.3] | 2.9 [2.3 to 3.8] | 2.3 [1.9 to 2.8] | 2.7 [2.0 to 3.6]
  Day 28 IgG to A/Victoria/361/2011 (H3N2) | 2.9 [2.3 to 3.6] | 3.5 [2.6 to 4.5] | 6.0 [4.5 to 7.8] | 7.7 [5.7 to 10.4]
  Day 0 IgG to B/Brisbane/60/2008 | 2.6 [2.0 to 3.2] | 2.6 [2.0 to 3.5] | 2.1 [1.8 to 2.4] | 2.4 [1.9 to 3.0]
  Day 28 IgG to B/Brisbane/60/2008 | 2.7 [2.2 to 3.4] | 2.9 [2.2 to 3.8] | 4.9 [3.7 to 6.3] | 4.2 [3.2 to 5.6]
  Day 0 IgG to B/Wisconsin/1/2010 | 1.7 [1.4 to 1.9] | 1.6 [1.3 to 1.8] | 1.5 [1.3 to 1.6] | 1.6 [1.3 to 1.9]
  Day 28 IgG to B/Wisconsin/1/2010 | 1.6 [1.4 to 1.9] | 1.6 [1.4 to 1.9] | 1.9 [1.6 to 2.2] | 5.0 [3.4 to 7.2]

6. Primary Outcome: Number of Infant Participants With Medically Attended Respiratory or Gastrointestinal AEs 28-42 Days After Maternal Vaccination
Description: Maternal participants were contacted by telephone at Day 42 to report all medically attended respiratory or gastrointestinal adverse events occurring in the infant participants between 28 and 42 days after maternal vaccination.
Time Frame: Within 28-42 days after maternal vaccination
Population: All infant participants for whom the maternal participants were contacted are included in the analysis population description. One maternal participant was not contacted.
Measure: Number; unit: participants
Arm/Group | Infant LAIV | Infant TIV
Number analyzed (Participants) | 124 | 125
participants
  Respiratory AE | 7 | 5
  Gastrointestinal AE | 2 | 0

7. Secondary Outcome: Geometric Mean Titers (GMT) in Maternal Sera of Hemagglutination Inhibition (HAI) Antibodies to Each of the Influenza Strains in the Vaccine Received
Description: Blood was collected for HAI assay at Day 0 prior to vaccination and again at 28 days following vaccination. The HAI assay was conducted with the antigens in the 2011-2012 seasonal influenza vaccine, A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008, those in the 2012-2013 seasonal influenza vaccine, A/Victoria/361/2011 and B/Wisconsin/1/2010, and the antigen in both seasons's vaccine, A/California/7/2009 (H1N1). The lower limit of detection for the assay was a titer of 10, sera samples below detection were given a value of 5 for analysis.
Time Frame: Day 0 and 28 post vaccination
Population: All enrolled maternal participants with results reported are included in this analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Maternal TIV 2011-2012 | Maternal TIV 2012-2013
Number analyzed (Participants) | 75 | 48 | 74 | 50
titer
  Day 0 - A/Perth/16/2009 (H3N2) | 45.5 [32.6 to 63.5] | 53.0 [36.1 to 77.8] | 32.9 [23.5 to 46.0] | 52.1 [37.7 to 71.9]
  Day 28 - A/Perth/16/2009 (H3N2) | 51.6 [37.2 to 71.5] | 59.9 [41.6 to 86.2] | 119.7 [88.2 to 162.4] | 133.6 [103.7 to 172.2]
  Day 0 - B/Brisbane/60/2008 | 20.2 [16.2 to 25.1] | 18.2 [14.2 to 23.4] | 15.7 [12.8 to 19.2] | 17.5 [14.1 to 21.8]
  Day 28 - B/Brisbane/60/2008 | 21.6 [17.4 to 26.9] | 18.5 [14.3 to 23.8] | 42.3 [33.1 to 54.1] | 31.0 [25.2 to 38.0]
  Day 0 - A/Victoria/361/2011 | 47.0 [33.2 to 66.6] | 60.4 [42.5 to 85.7] | 38.0 [26.6 to 54.2] | 62.8 [43.7 to 90.2]
  Day 28 - A/Victoria/361/2011 | 56.3 [39.7 to 79.8] | 81.2 [60.1 to 109.6] | 207.0 [161.1 to 265.9] | 247.6 [194.2 to 315.6]
  Day 0 - B/Wisconsin/1/2010 | 10.3 [8.4 to 12.7] | 8.7 [7.0 to 10.7] | 9.1 [7.6 to 11.0] | 10.6 [8.6 to 13.1]
  Day 28 - B/Wisconsin/1/2010 | 10.9 [8.9 to 13.4] | 9.0 [7.4 to 10.9] | 15.8 [12.6 to 19.9] | 41.1 [30.2 to 56.1]
  Day 0 -A/California/7/2009 (H1N1) | 44.7 [31.9 to 62.6] | 44.6 [31.6 to 63.0] | 42.9 [30.1 to 61.1] | 64.1 [43.1 to 95.3]
  Day 28 - A/California/7/2009 (H1N1) | 46.8 [33.6 to 65.1] | 44.9 [31.8 to 63.4] | 382.3 [284.3 to 514.2] | 197.0 [146.1 to 265.7]

8. Secondary Outcome: Number of Maternal Participants With Season-specific LAIV Influenza A and B Strains Detected in Respiratory Secretions Prior to Vaccination.
Description: Nasal swab samples were collected from all maternal participants prior to vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. The data coordinating center selected 25% of participants in the TIV group for testing to serve as an internal control for the assay.
Time Frame: Day 0 prior to vaccination
Population: All participants with samples selected for testing by the data coordinating center, 100% of LAIV recipients and 25% of TIV recipients, are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Maternal TIV 2011-2012 | Maternal TIV 2012-2013
Number analyzed (Participants) | 72 | 48 | 16 | 12
participants
  Influenza A - PCR negative, cell culture negative | 72 | 47 | 16 | 12
  Influenza A - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture negative | 0 | 1 | 0 | 0
  Influenza A - PCR positive, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR negative, cell culture negative | 72 | 48 | 16 | 12
  Influenza B - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture negative | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture positive | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Maternal Participants With Season-specific LAIV Influenza A and B Strains Detected in Respiratory Secretions at Day 2 Post Vaccination.
Description: Nasal swab samples were collected from all maternal participants at Day 2 post vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. The data coordinating center selected 25% of participants in the TIV group for testing to serve as an internal control for the assay.
Time Frame: Day 2 post vaccination
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Maternal TIV 2011-2012 | Maternal TIV 2012-2013
Number analyzed (Participants) | 73 | 47 | 19 | 12
participants
  Influenza A - PCR negative, cell culture negative | 51 | 41 | 19 | 12
  Influenza A - PCR negative, cell culture positive | 1 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture negative | 16 | 6 | 0 | 0
  Influenza A - PCR positive, cell culture positive | 5 | 0 | 0 | 0
  Influenza B - PCR negative, cell culture negative | 39 | 30 | 19 | 12
  Influenza B - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture negative | 21 | 13 | 0 | 0
  Influenza B - PCR positive, cell culture positive | 13 | 4 | 0 | 0

10. Primary Outcome: Number of Maternal Participants Reporting Fever After Vaccination
Description: Participants were provided with a thermometer and a memory aid on which to record daily oral temperatures for 8 days after vaccination (Day 0-7). The protocol defined fever as oral temperature of 37.8 degrees Celsius or higher. Participants are counted as experiencing fever if they reported oral temperatures of 37.8 degrees Celsius or higher on any of the 8 days.
Time Frame: Day 0-7 post vaccination
Population: All enrolled maternal participants are included in this analysis population.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV | Maternal TIV
Number analyzed (Participants) | 124 | 124
participants | 2 | 1

11. Primary Outcome: Number of Maternal Participants Reporting Solicited Subjective Systemic Symptoms After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, nausea, weakness, and chills for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 post vaccination
Population: All enrolled maternal participants are included in this analysis population.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV | Maternal TIV
Number analyzed (Participants) | 124 | 124
participants
  Feverishness | 7 | 6
  Malaise | 45 | 38
  Myalgia | 14 | 23
  Headache | 53 | 48
  Nausea | 5 | 9
  Weakness | 3 | 3
  Chills | 3 | 3

12. Primary Outcome: Number of Maternal Participants Reporting Solicited Subjective Local Symptoms After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of nasal congestion, runny nose, cough, sore throat, nasal bleeding, pain at injection site, tenderness at injection site, and swelling at injection site for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 post vaccination
Population: All enrolled maternal participants are included in this analysis population.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV | Maternal TIV
Number analyzed (Participants) | 124 | 124
participants
  Nasal congestion | 56 | 26
  Runny nose | 51 | 38
  Cough | 7 | 8
  Sore throat | 39 | 32
  Nasal bleeding | 3 | 1
  Pain at Injection Site | 9 | 70
  Tenderness at injection site | 17 | 100
  Swelling at injection site | 6 | 18

13. Primary Outcome: Number of Maternal Participants Reporting Solicited Quantitative Local Symptoms After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of redness and swelling for 8 days after vaccination (Day 0-7). If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Day 0-7 post vaccination
Population: All enrolled maternal participants are included in this analysis population.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV | Maternal TIV
Number analyzed (Participants) | 124 | 124
participants
  Redness | 13 | 23
  Swelling | 6 | 17

14. Secondary Outcome: Number of Maternal Participants With Season-specific LAIV Influenza A and B Strains Detected in Respiratory Secretions at Day 8 Post Vaccination.
Description: Nasal swab samples were collected from all maternal participants at Day 8 post vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. The data coordinating center selected 25% of participants in the TIV group for testing to serve as an internal control for the assay.
Time Frame: Day 8 post vaccination
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Maternal TIV 2011-2012 | Maternal TIV 2012-2013
Number analyzed (Participants) | 72 | 47 | 19 | 12
participants
  Influenza A - PCR negative, cell culture negative | 71 | 47 | 19 | 12
  Influenza A - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture negative | 1 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR negative, cell culture negative | 65 | 43 | 19 | 13
  Influenza B - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture negative | 6 | 2 | 0 | 0
  Influenza B - PCR positive, cell culture positive | 1 | 2 | 0 | 0

15. Secondary Outcome: Number of Infant Participants With Season-specific LAIV Influenza A and B Strains Detected in Respiratory Secretions Prior to Vaccination.
Description: Nasal swab samples were collected from all infant participants prior to vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. The data coordinating center selected 25% of participants in the TIV group for testing to serve as an internal control for the assay.
Time Frame: Day 0 prior to vaccination
Population: as for outcome 8
Measure: Number; unit: participants
Groups:
- Infant LAIV 2011-2012: Infants of women enrolled to receive LAIV in the 2011-2012 season were enrolled separately in the protocol to be followed for safety outcomes.
- Infant LAIV 2012-2013: Infants of women enrolled to receive LAIV in the 2012-2013 season were enrolled separately in the protocol to be followed for safety outcomes.
- Infant TIV 2011-2012: Infants of women enrolled to receive TIV in the 2011-2012 season were enrolled separately in the protocol to be followed for safety outcomes.
- Infant TIV 2012-2013: Infants of women enrolled to receive TIV in the 2012-2013 season were enrolled separately in the protocol to be followed for safety outcomes.
Arm/Group | Infant LAIV 2011-2012 | Infant LAIV 2012-2013 | Infant TIV 2011-2012 | Infant TIV 2012-2013
Number analyzed (Participants) | 71 | 48 | 19 | 13
participants
  Influenza A - PCR negative, cell culture negative | 71 | 48 | 19 | 13
  Influenza A - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture negative | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR negative, cell culture negative | 71 | 48 | 19 | 13
  Influenza B - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture negative | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture positive | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Infant Participants With Season-specific LAIV Influenza A and B Strains Detected in Respiratory Secretions at Day 2 Post Vaccination.
Description: Nasal swab samples were collected from all infant participants at Day 2 post vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. The data coordinating center selected 25% of participants in the TIV group for testing to serve as an internal control for the assay.
Time Frame: Day 2 post vaccination
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Infant LAIV 2011-2012 | Infant LAIV 2012-2013 | Infant TIV 2011-2012 | Infant TIV 2012-2013
Number analyzed (Participants) | 72 | 44 | 20 | 12
participants
  Influenza A - PCR negative, cell culture negative | 71 | 44 | 20 | 12
  Influenza A - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture negative | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture positive | 1 | 0 | 0 | 0
  Influenza B - PCR negative, cell culture negative | 72 | 44 | 20 | 12
  Influenza B - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture negative | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture positive | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Infant Participants With Season-specific LAIV Influenza A and B Strains Detected in Respiratory Secretions at Day 8 Post Vaccination.
Description: Nasal swab samples were collected from all infant participants at Day 8 post vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. The data coordinating center selected 25% of participants in the TIV group for testing to serve as an internal control for the assay.
Time Frame: Day 8 post vaccination
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Infant LAIV 2011-2012 | Infant LAIV 2012-2013 | Infant TIV 2011-2012 | Infant TIV 2012-2013
Number analyzed (Participants) | 72 | 47 | 19 | 13
participants
  Influenza A - PCR negative, cell culture negative | 72 | 47 | 19 | 13
  Influenza A - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture negative | 0 | 0 | 0 | 0
  Influenza A - PCR positive, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR negative, cell culture negative | 72 | 47 | 19 | 13
  Influenza B - PCR negative, cell culture positive | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture negative | 0 | 0 | 0 | 0
  Influenza B - PCR positive, cell culture positive | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Maternal Participants Positive for the Season-specific LAIV Influenza A Strain in Respiratory Secretions at Day 0 Who Were Positive for H1N1 and/or H3N2 Strains.
Description: Nasal swab samples were collected from all maternal participants prior to vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. Those who were positive for the Influenza A strain were further tested to identify the H1N1 and H3N2 strain.
Time Frame: Day 0 prior to vaccination
Population: The analysis population is limited to participants who were positive by PCR and/or cell culture for the vaccine strain of Influenza A.
Measure: Number; unit: participants
Arm/Group | Maternal LAIV 2012-2013
Number analyzed (Participants) | 1
participants
  H1N1 - PCR negative, cell culture negative | 1
  H1N1 - PCR negative, cell culture positive | 0
  H1N1 - PCR positive, cell culture negative | 0
  H1N1 - PCR positive, cell culture positive | 0
  H3N2 - PCR negative, cell culture negative | 1
  H3N2 - PCR negative, cell culture positive | 0
  H3N2 - PCR positive, cell culture negative | 0
  H3N2 - PCR positive, cell culture positive | 0

19. Secondary Outcome: Number of Maternal and Infant Participants Positive for the Season-specific LAIV Influenza A Strain in Respiratory Secretions at Day 2 Who Were Positive for H1N1 and/or H3N2 Strains.
Description: Nasal swab samples were collected from all maternal and infant participants at Day 2 post vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. Those who were positive for the Influenza A strain were further tested to identify the H1N1 and H3N2 strain.
Time Frame: Day 2 post vaccination
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Infant LAIV 2011-2012
Number analyzed (Participants) | 21 | 6 | 1
participants
  H1N1 - PCR negative, cell culture negative | 11 | 3 | 0
  H1N1 - PCR negative, cell culture positive | 4 | 0 | 1
  H1N1 - PCR positive, cell culture negative | 5 | 3 | 0
  H1N1 - PCR positive, cell culture positive | 1 | 0 | 0
  H3N2 - PCR negative, cell culture negative | 7 | 2 | 0
  H3N2 - PCR negative, cell culture positive | 0 | 0 | 0
  H3N2 - PCR positive, cell culture negative | 9 | 4 | 0
  H3N2 - PCR positive, cell culture positive | 5 | 0 | 1

20. Secondary Outcome: Number of Maternal Participants Positive for the Season-specific LAIV Influenza A Strain in Respiratory Secretions at Day 8 Who Were Positive for H1N1 and/or H3N2 Strains.
Description: Nasal swab samples were collected from all maternal participants at Day 8 post vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine in respiratory secretions. Those who were positive for the Influenza A strain were further tested to identify the H1N1 and H3N2 strain.
Time Frame: Day 8 post vaccination
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Maternal LAIV 2011-2012
Number analyzed (Participants) | 1
participants
  H1N1 - PCR negative, cell culture negative | 1
  H1N1 - PCR negative, cell culture positive | 0
  H1N1 - PCR positive, cell culture negative | 0
  H1N1 - PCR positive, cell culture positive | 0
  H3N2 - PCR negative, cell culture negative | 1
  H3N2 - PCR negative, cell culture positive | 0
  H3N2 - PCR positive, cell culture negative | 0
  H3N2 - PCR positive, cell culture positive | 0

21. Secondary Outcome: Number of Maternal Participants With Season-specific LAIV Influenza A and B Strains Detected in Breast Milk Following Vaccination.
Description: Breast milk was collected from all maternal participants prior at Days 2 and 8 post vaccination for PCR and cell culture to assess for the presence of the viruses in the LAIV vaccine. The data coordinating center selected 25% of participants in the TIV group for testing to serve as an internal control for the assay.
Time Frame: Day 2 and 8 post vaccination
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Maternal TIV 2011-2012 | Maternal TIV 2012-2013
Number analyzed (Participants) | 73 | 47 | 19 | 12
participants
  Day 2 - Influenza A | 0 | 0 | 0 | 0
  Day 8 - Influenza A | 0 | 0 | 0 | 0
  Day 2- Influenza B | 0 | 0 | 0 | 0
  Day 8 - Influenza B | 0 | 0 | 0 | 0

22. Secondary Outcome: ELISA IgA and IgG GMT to Each of the Influenza Strains in the Vaccine Received in Sera of Maternal Subjects
Description: Blood was collected from maternal subjects on Day 0 prior to vaccination, and at Day 28 post vaccination for assessment of IgA and IgG antibodies with a standard ELISA assay. The ELISA assay was conducted with the antigens in the 2011-2012 seasonal influenza vaccine, A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008, those in the 2012-2013 seasonal influenza vaccine, A/Victoria/361/2011 and B/Wisconsin/1/2010, and the antigen in both seasons' vaccines, A/California/7/2009 (H1N1). The lower limit of detection is 5.82 units/mL for IgA and 2.56 units/mL for IgG. Titers below the limit of detection were reported as one-half the limit of detection.
Time Frame: Day 0 and Day 28 post vaccination
Population: All enrolled maternal participants with results reported are included in this analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: units/mL
Arm/Group | Maternal LAIV 2011-2012 | Maternal LAIV 2012-2013 | Maternal TIV 2011-2012 | Maternal TIV 2012-2013
Number analyzed (Participants) | 75 | 48 | 74 | 50
units/mL
  Day 0 IgA to A/California/7/2009 (H1N1) | 180.3 [132.2 to 245.9] | 248.8 [163.4 to 378.6] | 220.0 [156.6 to 309.2] | 212.9 [140.7 to 322.1]
  Day 28 IgA to A/California/7/2009 (H1N1) | 211.0 [152.5 to 291.9] | 281.0 [193.6 to 407.8] | 845.3 [559.9 to 1276.2] | 417.2 [273.9 to 635.4]
  Day 0 IgA to A/Perth/16/2009 (H3N2) | 724.2 [527.3 to 994.6] | 1065.7 [734.4 to 1546.5] | 611.2 [466.1 to 801.5] | 697.7 [512.0 to 950.8]
  Day 28 IgA to A/Perth/16/2009 (H3N2) | 949.6 [690.2 to 1306.5] | 1400.9 [1010.8 to 1941.5] | 1514.9 [1154.3 to 1988.3] | 1262.5 [913.4 to 1745.1]
  Day 0 IgA to A/Victoria/361/2011 (H3N2) | 697.7 [509.7 to 955.1] | 986.4 [685.6 to 1419.2] | 601.9 [457.9 to 791.1] | 678.2 [491.7 to 935.6]
  Day 28 IgA to A/Victoria/361/2011 (H3N2) | 920.1 [669.7 to 1264.1] | 1308.8 [949.5 to 1804.0] | 1455.3 [1103.2 to 1919.6] | 1206.2 [875.5 to 1661.9]
  Day 0 IgA to B/Brisbane/60/2008 | 459.4 [361.9 to 583.1] | 632.6 [440.0 to 909.7] | 408.3 [310.6 to 536.7] | 532.1 [376.2 to 752.7]
  Day 28 IgA to B/Brisbane/60/2008 | 637.2 [505.9 to 802.7] | 745.8 [510.8 to 1089.1] | 753.0 [561.9 to 1009.2] | 933.4 [648.0 to 1344.6]
  Day 0 IgA to B/Wisconsin/1/2010 | 217.5 [172.2 to 274.7] | 264.9 [183.3 to 382.7] | 228.3 [176.1 to 295.9] | 276.4 [196.1 to 389.4]
  Day 28 IgA to B/Wisconsin/1/2010 | 281.3 [226.8 to 348.9] | 382.0 [265.0 to 550.6] | 314.1 [241.5 to 408.5] | 1034.3 [625.1 to 1711.3]
  Day 0 IgG to A/California/7/2009 (H1N1) | 1224.8 [988.8 to 1517.1] | 1014.6 [764.2 to 1347.0] | 1133.5 [876.4 to 1465.9] | 1301.6 [964.9 to 1755.7]
  Day 28 IgG to A/California/7/2009 (H1N1) | 1193.9 [963.1 to 1479.9] | 1078.9 [823.0 to 1414.5] | 5834.1 [4507.4 to 7551.4] | 3526.6 [2794.0 to 4451.3]
  Day 0 IgG to A/Perth/16/2009 (H3N2) | 2228.8 [1790.2 to 2774.8] | 2022.0 [1557.9 to 2624.2] | 1798.5 [1375.6 to 2351.5] | 2244.7 [1775.8 to 2837.4]
  Day 28 IgG to A/Perth/16/2009 (H3N2) | 2389.8 [1931.9 to 2956.2] | 2296.1 [1780.8 to 2960.4] | 5594.7 [4546.6 to 6884.5] | 5655.1 [4556.8 to 7018.0]
  Day 0 IgG to A/Victoria/361/2011 (H3N2) | 2496.3 [1998.8 to 3117.7] | 2065.7 [1537.6 to 2775.2] | 2018.9 [1566.0 to 2602.8] | 2242.8 [1724.4 to 2917.1]
  Day 28 IgG to A/Victoria/361/2011 (H3N2) | 2742.3 [2217.6 to 3391.3] | 2275.6 [1697.7 to 3050.3] | 6132.1 [4993.7 to 7530.0] | 5996.0 [4676.6 to 7687.7]
  Day 0 IgG to B/Brisbane/60/2008 | 2844.8 [2240.9 to 3611.4] | 2225.8 [1630.4 to 3038.7] | 2159.5 [1716.8 to 2716.2] | 2617.4 [2069.6 to 3310.3]
  Day 28 IgG to B/Brisbane/60/2008 | 3064.5 [2465.3 to 3809.3] | 2381.0 [1760.7 to 3219.9] | 5813.6 [4851.7 to 6966.1] | 3897.7 [3149.6 to 4823.5]
  Day 0 IgG to B/Wisconsin/1/2010 | 1279.6 [988.2 to 1656.8] | 919.4 [652.0 to 1296.5] | 1071.2 [840.9 to 1364.6] | 1532.9 [1146.3 to 2049.9]
  Day 28 IgG to B/Wisconsin/1/2010 | 1337.2 [1048.0 to 1706.4] | 1185.2 [868.5 to 1617.3] | 1914.0 [1586.3 to 2309.3] | 5840.2 [4417.0 to 7722.0]

ADVERSE EVENTS:
Time Frame: Solicited systemic and local symptoms were collected for 8 days after vaccination (maternal), 10 days (infant). Unsolicited AEs were collected for 28 days and SAEs and new onset chronic medical conditions were collected for 6 months after vaccination.
Description: For events solicited on the Memory Aid, a participant was considered to have 1 event if it was reported as experienced at any time in the 8 day period for maternal arms, 10 days for infant arms. Number at risk is 0 for infant arms for events solicited only for maternal arms, and 0 for maternal arms for events solicited only for infants.
Arm/Group | Maternal LAIV | Maternal TIV | Infant LAIV | Infant TIV
Serious Adverse Events (participants affected / at risk) | 1/124 | 0/124 | 2/124 | 1/125
Other Adverse Events (participants affected / at risk) | 106/124 | 122/124 | 102/124 | 101/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal LAIV (N=124) | Maternal TIV (N=124) | Infant LAIV (N=124) | Infant TIV (N=125)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital syphilis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Maternal LAIV (N=124) | Maternal TIV (N=124) | Infant LAIV (N=124) | Infant TIV (N=125)
Feeling hot (General disorders) | 7 (7) | 6 (6) | 0/0 (0) | 0/0 (0) — Solicited as 'feverishness' on the memory aid
Malaise (General disorders) | 45 (45) | 38 (38) | 0/0 (0) | 0/0 (0) — Solicited at 'fatigue/malaise' on the memory aid
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 23 (23) | 0/0 (0) | 0/0 (0) — Solicited as 'generalized body aches/myalgia' on the memory aid
Headache (Nervous system disorders) | 53 (53) | 48 (48) | 0/0 (0) | 0/0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 9 (9) | 0/0 (0) | 0/0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 56 (56) | 26 (26) | 54 (54) | 54 (54)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 51 (51) | 38 (38) | 18 (18) | 30 (30) — Solicited as 'runny nose' on the memory aid
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8) | 15 (15) | 18 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 39 (39) | 32 (32) | 0/0 (0) | 0/0 (0) — Solicited as 'sore throat' on the memory aid
Injection site pain (General disorders) | 9 (9) | 70 (70) | 0/0 (0) | 0/0 (0)
Tenderness (General disorders) | 17 (17) | 100 (100) | 0/0 (0) | 0/0 (0) — Solicited specifically for at the injection site on the memory aid.
Injection site erythema (General disorders) | 13 (13) | 23 (23) | 0/0 (0) | 0/0 (0)
Injection site swelling (General disorders) | 6 (6) | 18 (18) | 0/0 (0) | 0/0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 13 (13) | 15 (15) | 10 (10)
Irritability (General disorders) | 0 (0) | 0 (0) | 5 (5) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 7 (7)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 28 (28) | 23 (23)
Somnolence (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 42 (42) | 33 (33) — Solicited as 'drowsiness' on the memory aid.
Irritability (General disorders) | 0/0 (0) | 0/0 (0) | 74 (74) | 56 (56) — Solicited as 'irritability/fussiness' on the memory aid
Decreased appetite (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 20 (20) | 14 (14) — Solicited as 'loss of appetite' on the memory aid
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 12 (12) | 7 (7) — Solicited as 'difficulty breathing' on the memory aid

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less